CLINICAL TRIAL: NCT02459561
Title: A Randomised Controlled Trial of a Duodenal Sleeve Bypass Device (EndoBarrier)Compared With Standard Medical Therapy for the Management of Obese Subjects With Type 2 Diabetes
Brief Title: EndoBarrier TM Gastrointestinal Liner Diabetes Trial
Acronym: EndoBarrier
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Imperial College London (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); University Hospital Southampton NHS Foundation Trust (Other); Brunel University (Other); University of Surrey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14SM2015
Record Dates: First submitted 2015-05-20; First posted 2015-06-02 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Overweight and Obesity; Diabetes
Keywords: Obesity; Diabetes; Overweight; Medical device; Endobarrier; Clinical trial; Diet; Exercise; Body weight; Medical therapy; Medicine; Device; Randomised; Control; Intervention; EndoBarrier Medical device
MeSH Terms: conditions — Overweight; Obesity; Diabetes Mellitus; Motor Activity; Body Weight

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EndoBarrier Arm (Experimental): The EndoBarrier Gastrointestinal Liner device received CE Mark for 12 months implant duration on 11 December 2009 and is a single use, minimally invasive device, used to achieve weight loss and improve Type 2 Diabetes status in subjects who are obese. The intent of the EndoBarrier Gastrointestinal Liner is to mimic portions of the standard Roux-en-Y bypass procedure. The device consists of 3 components: the implant, the delivery system, and the removal system. At study visit 4, after eight hours fasting, 80 subjects will arrive to the pre- assessment unit as part of the theatres at St. Mary's Hospital or Southampton Hospital and receive the EndoBarrier TM Gastrointestinal Liner as part of the EndoBarrier Arm Intervention.
  Interventions: Device: EndoBarrier TM Gastrointestinal Liner
- Medical Therapy Arm (Other): The standard medical therapy arm will be carried out in accordance with the guidelines of the American Diabetes Association. These guidelines have been chosen as they are applicable to an International audience and thus would adhere to the current best worldwide practice that would still be likely to be relevant when the results are published following study completion.
  Diabetes reviews appointments with a Diabetologist/Endocrinologist will be performed with the control arm patients at visits 2, 4, 6, 7, 9, 11, 12, 13 and 15.
  At study visit 4, 80 subjects will arrive at Mary's Hospital or Southampton Hospital and receive the best Medical Care and dietary advice as part of the Medical Therapy Arm Interventions.
  Interventions: Other: Best Medical Care

INTERVENTIONS:
Device: EndoBarrier TM Gastrointestinal Liner — If subjects are randomised into the EndoBarrier Group of the trial they will receive the device for 12 months followed a 12 months follow-up period.
  Arms: EndoBarrier Arm
Other: Best Medical Care — If subjects are randomised into the Control Group of the trial they will receive best medical care and dietitian advice for 12 months followed a 12 months follow-up period.
  Arms: Medical Therapy Arm

SUMMARY:
The management of obesity is challenging and obesity surgery is by far the most effective treatment currently available. Recent medical research indicates that it also improves the management of blood glucose levels in people with type 2 diabetes. Obesity surgery carries different risks and benefits and it is important to balance these by choosing the right procedure for each patient. Therefore new effective strategies to prevent and reduce obesity and its complications such as type 2 diabetes mellitus are needed. This study is designed to see whether a new device called the EndoBarrier Gastrointestinal Liner helps patients manage their blood sugar levels and lose weight. It is a randomised, placebo controlled trial which compares the potential of the EndoBarrier device with conventional drug therapy, diet and exercise for obesity related type 2 diabetes, and their effectiveness on metabolic state (HbA1c reduced by 20% and blood pressure below 135/85), weight loss, and quality of life. It will further evaluate whether any other conditions that may be related to obesity could become less severe and collect information about complications to determine the safety of the device. The study will also perform various measurements and tests to understand the underlying mechanism of the device. After an initial screening visit to determine patients eligibility, they will be invited for 14 subsequent visits. Patients will be randomised into either having the EndoBarrier device or standard medical therapy treatment for 12 months followed by another 12 months follow-up period. They will also be routinely seen by specialist dietitian who will provide dietetic support throughout the study.

DETAILED DESCRIPTION:
Patients will be recruited via primary care and secondary care trusts. After an initial screening visit to determine subject's eligibility, they will be randomised to either the EndoBarrier or Control arm (conventional medical therapy including dietary counselling), and invited for 15 study visits over 24 months. The standard medical therapy drug titrations will be carried out in accordance with the guidelines of the American Diabetes Association. These guidelines have been chosen as they are applicable to an International audience and thus would adhere to the current best worldwide practice that would still be likely to be relevant when the results of this trial are published following study completion.

Patients will receive the intervention for 12 months and then be followed up for 12 months. They will be contacted via telephone in between visits to monitor any problems and boost motivation.

The main outcome of this study is to compare the EndoBarrier device with conventional medical therapy, diet and exercise for obesity related type 2 diabetes and their effectiveness on:

1. Metabolic state as defined by the International Diabetes Federation (IDF) with an HbA1c < 6% (or < 42 mmol/mol) and a blood pressure < 135/85mmHg
2. Absolute weight loss.

Patients will also be invited to participate in one of 3 sub-groups as part of the mechanistic studies (Group 1: functional MRI (fMRI), Group 2: insulin clamps or Group 3: food preference). Participation in the sub-studies is optional.

The following assessments will be performed at visit 1 (Screening Visit):

Informed consent, inclusion and exclusion criteria, demographics, medical history, physical examination, body measurements including height, weight and waist , vital signs, ECG, urine albumin-creatinine ratio, routine haematology and biochemistry, C13 urea breath test and urine pregnancy test, if applicable. Additional checks will be completed if the subject consents to take part in a sub-group mechanistic study.

Once all data including blood test results related to the screening have been obtained, the Investigator will review the subject's eligibility to continue in the trial. If the subject is eligible after this review, the subject will be randomised into one of the two study arms (EndoBarrier or Control).

Both groups will undergo the following measurements:

* Body weight and waist circumference, blood pressure, changes in illness and medication and adverse events will be checked at all visits.
* Blood samples will be obtained at 13 visits
* Urine albumin:creatinine ratio: urine samples will be collected at visit 3, 5, 8, 10 and 14
* Questionnaires (Health Economics) will be completed at visits 3, 5, 6, 7, 8, 10 and 14.
* Dietary counselling: at visits 2, 4 (control arm only), 6, 7, 9, 11, 12, 13, and 15 subjects will receive diet (either in groups or individually) by a qualified dietitian.

EndoBarrier group:

Visit 2 (- 4 weeks) will include dietary counselling with a dietitian, dietary preparation pre- and post-intervention and a medical consultation (including distribution of proton pump inhibitors) in preparation for the EndoBarrier implant.

At visit 4 (0 weeks) the EndoBarrier device will be implanted. The subject will attended the hospital in a fasting state and will receive a general anaesthetic before the device placement procedure. A small tube (the endoscope) is inserted into the mouth and guided to the small intestine for visual examination of this area by the physician. Then a guide wire will be inserted through the endoscope, after which the endoscope is removed but the guide wire is left in place. A capsule (containing the device) is placed on the guide wire and guided to the destination in the small intestine. The physician can see the capsule under x-rays as it is moved towards the small intestine. When the physician determines that the capsule has reached the correct location, the guide wire is removed, which releases the device. When the device is released, it also releases a small plastic ball (slightly larger than a pea). The ball is excreted naturally via a stool. Normally, this does not cause any discomfort. The device remains in the small intestine until it is removed after 12 months.

After the procedure (up to 12 hours) the subject may need to stay overnight in the hospital so the physician can monitor their condition, but this usually is not required.

During insertion fluroscopy will be used to determine the position of the device. Videos and photos of the fluoroscopy images are recorded to help the investigators make treatment decisions and may be passed on to the study sponsor. The images will not contain any patient identifiable data but will be labelled with initials and study participation number only.

At visit 11 (12 months) the EndoBarrier device will be removed. The removal procedure is comparable to the placement procedure but usually requires less time. Before the device removal procedure, the subject will receive a general anaesthetic. During device removal, an endoscope is inserted into the mouth and guided to the small intestine for visual examination of this area by the physician. A guide wire is inserted into the endoscope. The end of the endoscope has a small hook, which the physician will use to pull the device back into the endoscope. The endoscope containing the device is then removed through the mouth. The physician will then insert the endoscope again to inspect the area where the device was placed. After the procedure, the subject can return home.

All subjects in the EndoBarrier arm will see a gastroenterologist or equivalent specialist at study visit 2, 6, 7, 9, 11, 12, 13 and 15 to discuss their well-being and any questions regarding their EndoBarrier implant. EndoBarrier patients will also receive frequent reviews with a diabetes specialist to review their medication regimen (visits 2, 6, 7, 9, 12, 13 and 15).

Control group (Standard Medical Therapy) Standard medical therapy will be carried out in accordance with the guidelines of the American Diabetes Association. Patients will be seen at visits 2, 4, 6, 7, 9, 11, 12, 13 and 15 for follow-up of their diabetes control by a diabetes specialist.

Both groups will provide a blood sample for DNA/RNA sampling: at visit 3 and samples for metabolomics (blood, urine, feces): at visits 3, 5, 8, 10 and 14

Subjects who agree to participate in a sub-study will be asked to complete additional tests including:

* Fasting Gut hormones and metabolites (Group 1-3): at visits 3, 5, 8, 10 and 14
* Post meal gut hormones and metabolites (Group 1 and 3): at visits 3, 5, 8, 10
* Eating and behaviour questionnaires (Group 1-3): at visits 3, 8, 10 and 14
* Functional MRI (Group 1): at visits 3 and 8
* Taste and Food preference (Group 3): at visits 3, 5, and 8
* Eating behaviour computerised tasks (Group 1 and 3): at visits 3, 8, 10 and 14
* Cognitive Assessment tasks (Group 1): at visits 3, 8 and 10
* Insulin Clamps (Group 2): at visits 3, 5, and 8

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years (male or female)
2. T2DM for at least 1 year (HbA1c 7.5-10.0% = 58-86 mmol/mol)
3. On oral T2DM medications (metformin is allowed, but not required)
4. BMI 30-50 kg/m2 with adequate insulin reserve as indicated with insulin C-peptide levels > 1665 pmol/L

Exclusion Criteria:

1. Language barrier, mental incapacity, unwillingness or inability to understand and be able to complete questionnaires
2. Non-compliance with eligibility criteria
3. Females of childbearing potential who are pregnant, breast-feeding or intend to become pregnant or are not using adequate or reliable contraceptive methods
4. Current use of insulin
5. Previous diagnosis with Type 1 DM or a history of ketoacidosis
6. Requirement of NSAIDs (non-steroidal anti-inflammatory drugs) or prescription of anticoagulation therapy during the implant period
7. History of iron deficiency and/or iron deficiency anaemia
8. Symptomatic gallstones or kidney stones at the time of screening
9. History of coagulopathy, upper gastro-intestinal bleeding conditions such as oesophageal or gastric varices, congenital or acquired intestinal telangiectasia
10. Previous GI surgery that could affect the ability to place the device or the function of the implant
11. History or presence of active H. pylori (if subjects are randomised into the EndoBarrier arm and have a history or presence of active H. pylori - tested during study visit 2 - they can receive appropriate treatment and then subsequently enrol into the study)
12. Family history of a known diagnosis or pre-existing symptoms of systemic lupus erythematosus, scleroderma or other autoimmune connective tissue disorder
13. Severe liver (AST, ALT or gGT >4 times upper limit) or kidney failure (serum creatinine >180mmol/l), estimated Glomerular Filtration Rate (GFR) cut-off is 60
14. Severe depression, unstable emotional or psychological characteristics (indicated by Beck Depression Inventory II score >28)
15. Poor dentition and inability to adequately chew food
16. Planned holidays up to three months following the EndoBarrier Implant
17. Previous EndoBarrier implantation
18. Metal implant unsuitable for MRI scanning and claustrophobia as contraindications for MRI scans (sub-group 1 - fMRI study only)
19. Vegetarian, vegan, gluten or lactose intolerance as unsuitable for fMRI food picture paradigm (sub-group 1 - fMRI only)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2018-10-18 (Actual); Study Completion 2019-05-15 (Estimated)

PRIMARY OUTCOMES:
HbA1c reduced by 20% | 2 years
  To compare the EndoBarrier with conventional medical therapy, diet and exercise for obesity related type II diabetes and their effectiveness on metabolic state as defined by the International Diabetes Federation (IDF) with an HbA1c reduced by 20%.

SECONDARY OUTCOMES:
HbA1c < 6% ( or < 42 mmol/mol) | 2 years
  HbA1c < 42 mmol/mol
Blood pressure < 135/85 | 2 years
  Blood pressure < 135/85
Absolute weight loss | 2 years
  Absolute weight loss
Changes in gut hormones before and after the EndoBarrier device | 2 years
  To investigate the mechanism of the effect of the EndoBarrier, venous blood samples will be taken at intervals by venepuncture through a cannula placed in the antecubital fossa. Serial plasma levels of glucose and other metabolites, bile acids, glucose, insulin, leptin, gut hormones (including ghrelin, GLP-1, PYY), adipocytokines and markers of insulin resistance, and inflammation will be measured. Assays will be performed by the Dept. of Chemical Pathology at Imperial College Healthcare NHS Trust and by in-house assays, outside contracts and commercial kits for radio-immunoassay and ELISA. These will be measured in the fasted and/or postprandial state for each patient and compared within and between the groups using parametric/non-parametric repeated measures statistical testing. Regressions will be performed with clinical outcomes (i.e. BMI, glucose control) to identify predictive markers and generate mechanistic hypotheses.
Changes in gut microbiome before and after the EndoBarrier device to investigate the mechanism of the effect of the EndoBarrier. | 2 years
  To investigate the mechanism of the effect of the EndoBarrier, plasma, urine and faecal samples for metabolomics will be collected at visit 3, 5, 8 and 10 and 14. All samples will be analysed using Mass spectroscopy and NMR spectroscopy. Metabolic datasets will be analysed using principal component analysis (PCA) and orthogonal partial least-squares analysis (O-PLS). The metabolic and microbial data will also be analysed in relation to response measurements such as BMI, gut hormone levels and etc. using O-PLS regression analysis and Bayesian approaches. A range of statistical methods will be optimised and applied to the data to identify weight loss and T2DM-associated microbiota and metabolites.
Changes in brain reward systems before and after the EndoBarrier device to investigate the mechanism of the effect of the EndoBarrier. | 2 years
  Patients will have fMRI scans to examine between brain function related to food reward and addictive behaviours at baseline and early after intervention, and these will be correlated to psychological questionnaires, computerised tasks, and test meals. Comparison of brain activation during fMRI paradigms and outcomes from behavioural measures of food hedonics and questionnaires will be compared between groups using a 2x2 ANOVA design including group (control vs. Endobarrier) between subject factor, time (baseline vs. follow-up visit) within subject factor, and group x time interaction to identify differential effects between groups. In addition linear regression will be performed to measure the correlation of variables at baseline or during the intervention with primary outcomes at 1 year e.g. weight loss and decreases in HbA1c within each group.
Changes in body fat content before and after the EndoBarrier device to investigate the mechanism of the effect of the EndoBarrier. | 2 years
  As well as baseline anthropometric measurements of height, weight, waist and hip circumference, patients will also have their percentage body fat determined by bio-electrical impedance analysis. This is a painless, safe procedure to measure total body fat involves lying on a bed, having two sticky pads placed on a hand and foot, and lying still for 1 minute, or standing on a metal platform for 1 minute so that the body's electrical resistance can be measured.
Changes in food preference before and after the EndoBarrier device to investigate the mechanism of the effect of the EndoBarrier. | 2 years
  Sweet taste detection testing: 7 ascending sucrose concentrations in solution will used to determine sweet detection thresholds. The subjects will sample the stimulus in the mouth and then spit the sample in a container to then indicate whether the stimulus was water or not. Consummatory taste reward: 5 ascending fat and sucrose solutions/ice-cream will be used to test responses in intensity ratings and hedonic reward. Participants will be asked to put the solutions into their mouths and then to spit it out into a bucket. While the solution is in the participants' mouths they will be asked to rate its intensity and pleasantness using visual analogue scales. Analysis: Sweet taste detection thresholds and visual analogue taste ratings will be quantified for each patient and compared within and between the groups at 3 time points using parametric/non-parametric repeated measures statistical testing.
Changes in biomarkers such as genetic markers before and after the EndoBarrier device | 2 years
  To investigate the mechanism of the effect of the EndoBarrier, blood (15 ml) will be taken to extract DNA and RNA for examination of genetic markers which predict weight loss, genetic abnormalities causing or contributing to obesity and insulin resistance (including array comparative genomic hybridization for copy number variations, epigenetic analysis, whole genome or exome sequencing, DNA sequencing of candidate genes (such as MC4R, POMC, leptin receptor, SIM1); and polymorphisms or mutations associated with obesity, diabetes mellitus, PCOS, fat distribution and body composition (using PCR based SNP analysis)56-58. RNA will be extracted from blood to perform genome-wide expression analysis.
Changes in hepatic or peripheral insulin sensitivity before and after the EndoBarrier device to investigate the mechanism of the effect of the EndoBarrier | 2 years
  Patients will undergo a euglycaemic hyperinsulinaemic clamp with stable isotope infusion to determine overall insulin and compartment-specific insulin sensitivity (liver, muscle and adipose depot). Blood samples will be taken every 5 minutes to measure blood glucose concentration and the dextrose infusion will be adjusted accordingly. Overall and tissue specific insulin sensitivity will be quantified for each patient and compared within and between the groups at 3 time points using parametric/non-parametric repeated measures statistical testing. Regressions will be performed with clinical outcomes (i.e. BMI, glucose control) to identify predictive markers and generate mechanistic hypotheses.
To estimate the cost-effectiveness of the EndoBarrier device compared with conventional treatment. | 2 years
  To estimate the cost-effectiveness of the EndoBarrier device compared with conventional treatment over the trial period using Quality of Life questionnaires. These comprise the EQ-5D-5L questionnaire to assess health-related quality of life, and a bespoke questionnaire designed to collect information about patients' use of health and social care resources (for costing purposes). The resource use questionnaire has been adapted from existing instruments and will ask patients to specify what services they have used since the previous assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Julian Teare, Professor, Principal Investigator — Imperial College London
Locations (1):
- Imperial Clinical Trials Unit, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Laferrere B, Swerdlow N, Bawa B, Arias S, Bose M, Olivan B, Teixeira J, McGinty J, Rother KI. Rise of oxyntomodulin in response to oral glucose after gastric bypass surgery in patients with type 2 diabetes. J Clin Endocrinol Metab. 2010 Aug;95(8):4072-6. doi: 10.1210/jc.2009-2767. Epub 2010 May 25. PMID 20501690
- [Background] Rubino F, Forgione A, Cummings DE, Vix M, Gnuli D, Mingrone G, Castagneto M, Marescaux J. The mechanism of diabetes control after gastrointestinal bypass surgery reveals a role of the proximal small intestine in the pathophysiology of type 2 diabetes. Ann Surg. 2006 Nov;244(5):741-9. doi: 10.1097/01.sla.0000224726.61448.1b. PMID 17060767
- [Background] Fairburn CG, Beglin SJ. Assessment of eating disorders: interview or self-report questionnaire? Int J Eat Disord. 1994 Dec;16(4):363-70. PMID 7866415
- [Background] Carver, C.S. & White, T.L. Behavioral-Inhibition, Behavioral Activation, and Affective Responses to Impending Reward and Punishment - the Bis Bas Scales. J Pers Soc Psychol 67, 319-333 (1994).
- [Background] Beck, A.T., Steer, R.A. & Brown, G.K. BDI-II, Beck depression inventory manual, (Psychological Corp, San Antonio, Tex, 1996).
- [Background] Horn NR, Dolan M, Elliott R, Deakin JF, Woodruff PW. Response inhibition and impulsivity: an fMRI study. Neuropsychologia. 2003;41(14):1959-66. doi: 10.1016/s0028-3932(03)00077-0. PMID 14572528
- [Result] Centers for Disease Control and Prevention (CDC). Prevalence of overweight and obesity among adults with diagnosed diabetes--United States, 1988-1994 and 1999-2002. MMWR Morb Mortal Wkly Rep. 2004 Nov 19;53(45):1066-8. PMID 15549021
- [Result] Hoerger TJ, Segel JE, Gregg EW, Saaddine JB. Is glycemic control improving in U.S. adults? Diabetes Care. 2008 Jan;31(1):81-6. doi: 10.2337/dc07-1572. Epub 2007 Oct 12. PMID 17934153
- [Result] Sjostrom L, Peltonen M, Jacobson P, Sjostrom CD, Karason K, Wedel H, Ahlin S, Anveden A, Bengtsson C, Bergmark G, Bouchard C, Carlsson B, Dahlgren S, Karlsson J, Lindroos AK, Lonroth H, Narbro K, Naslund I, Olbers T, Svensson PA, Carlsson LM. Bariatric surgery and long-term cardiovascular events. JAMA. 2012 Jan 4;307(1):56-65. doi: 10.1001/jama.2011.1914. PMID 22215166
- [Result] Mingrone G, Panunzi S, De Gaetano A, Guidone C, Iaconelli A, Leccesi L, Nanni G, Pomp A, Castagneto M, Ghirlanda G, Rubino F. Bariatric surgery versus conventional medical therapy for type 2 diabetes. N Engl J Med. 2012 Apr 26;366(17):1577-85. doi: 10.1056/NEJMoa1200111. Epub 2012 Mar 26. PMID 22449317
- [Result] Schauer PR, Kashyap SR, Wolski K, Brethauer SA, Kirwan JP, Pothier CE, Thomas S, Abood B, Nissen SE, Bhatt DL. Bariatric surgery versus intensive medical therapy in obese patients with diabetes. N Engl J Med. 2012 Apr 26;366(17):1567-76. doi: 10.1056/NEJMoa1200225. Epub 2012 Mar 26. PMID 22449319
- [Result] Dixon JB, le Roux CW, Rubino F, Zimmet P. Bariatric surgery for type 2 diabetes. Lancet. 2012 Jun 16;379(9833):2300-11. doi: 10.1016/S0140-6736(12)60401-2. Epub 2012 Jun 9. PMID 22683132
- [Result] le Roux CW, Aylwin SJ, Batterham RL, Borg CM, Coyle F, Prasad V, Shurey S, Ghatei MA, Patel AG, Bloom SR. Gut hormone profiles following bariatric surgery favor an anorectic state, facilitate weight loss, and improve metabolic parameters. Ann Surg. 2006 Jan;243(1):108-14. doi: 10.1097/01.sla.0000183349.16877.84. PMID 16371744
- [Result] Simonen M, Dali-Youcef N, Kaminska D, Venesmaa S, Kakela P, Paakkonen M, Hallikainen M, Kolehmainen M, Uusitupa M, Moilanen L, Laakso M, Gylling H, Patti ME, Auwerx J, Pihlajamaki J. Conjugated bile acids associate with altered rates of glucose and lipid oxidation after Roux-en-Y gastric bypass. Obes Surg. 2012 Sep;22(9):1473-80. doi: 10.1007/s11695-012-0673-5. PMID 22638681
- [Result] Patti ME, Houten SM, Bianco AC, Bernier R, Larsen PR, Holst JJ, Badman MK, Maratos-Flier E, Mun EC, Pihlajamaki J, Auwerx J, Goldfine AB. Serum bile acids are higher in humans with prior gastric bypass: potential contribution to improved glucose and lipid metabolism. Obesity (Silver Spring). 2009 Sep;17(9):1671-7. doi: 10.1038/oby.2009.102. Epub 2009 Apr 9. PMID 19360006
- [Result] Scholtz S, Miras AD, Chhina N, Prechtl CG, Sleeth ML, Daud NM, Ismail NA, Durighel G, Ahmed AR, Olbers T, Vincent RP, Alaghband-Zadeh J, Ghatei MA, Waldman AD, Frost GS, Bell JD, le Roux CW, Goldstone AP. Obese patients after gastric bypass surgery have lower brain-hedonic responses to food than after gastric banding. Gut. 2014 Jun;63(6):891-902. doi: 10.1136/gutjnl-2013-305008. Epub 2013 Aug 20. PMID 23964100
- [Result] Miras AD, Jackson RN, Jackson SN, Goldstone AP, Olbers T, Hackenberg T, Spector AC, le Roux CW. Gastric bypass surgery for obesity decreases the reward value of a sweet-fat stimulus as assessed in a progressive ratio task. Am J Clin Nutr. 2012 Sep;96(3):467-73. doi: 10.3945/ajcn.112.036921. Epub 2012 Jul 25. PMID 22836034
- [Result] Pournaras DJ, Osborne A, Hawkins SC, Vincent RP, Mahon D, Ewings P, Ghatei MA, Bloom SR, Welbourn R, le Roux CW. Remission of type 2 diabetes after gastric bypass and banding: mechanisms and 2 year outcomes. Ann Surg. 2010 Dec;252(6):966-71. doi: 10.1097/SLA.0b013e3181efc49a. PMID 21107106
- [Result] Rubino F, Schauer PR, Kaplan LM, Cummings DE. Metabolic surgery to treat type 2 diabetes: clinical outcomes and mechanisms of action. Annu Rev Med. 2010;61:393-411. doi: 10.1146/annurev.med.051308.105148. PMID 20059345
- [Result] Tarnoff M, Shikora S, Lembo A, Gersin K. Chronic in-vivo experience with an endoscopically delivered and retrieved duodenal-jejunal bypass sleeve in a porcine model. Surg Endosc. 2008 Apr;22(4):1023-8. doi: 10.1007/s00464-007-9652-7. Epub 2007 Nov 20. PMID 18030524
- [Result] Gersin KS, Keller JE, Stefanidis D, Simms CS, Abraham DD, Deal SE, Kuwada TS, Heniford BT. Duodenal- jejunal bypass sleeve: a totally endoscopic device for the treatment of morbid obesity. Surg Innov. 2007 Dec;14(4):275-8. doi: 10.1177/1553350607312901. PMID 18178916
- [Result] Sugerman HJ, Wolfe LG, Sica DA, Clore JN. Diabetes and hypertension in severe obesity and effects of gastric bypass-induced weight loss. Ann Surg. 2003 Jun;237(6):751-6; discussion 757-8. doi: 10.1097/01.SLA.0000071560.76194.11. PMID 12796570
- [Result] Rodriguez-Grunert L, Galvao Neto MP, Alamo M, Ramos AC, Baez PB, Tarnoff M. First human experience with endoscopically delivered and retrieved duodenal-jejunal bypass sleeve. Surg Obes Relat Dis. 2008 Jan-Feb;4(1):55-9. doi: 10.1016/j.soard.2007.07.012. PMID 18201671
- [Result] Gersin KS, Rothstein RI, Rosenthal RJ, Stefanidis D, Deal SE, Kuwada TS, Laycock W, Adrales G, Vassiliou M, Szomstein S, Heller S, Joyce AM, Heiss F, Nepomnayshy D. Open-label, sham-controlled trial of an endoscopic duodenojejunal bypass liner for preoperative weight loss in bariatric surgery candidates. Gastrointest Endosc. 2010 May;71(6):976-82. doi: 10.1016/j.gie.2009.11.051. Epub 2010 Mar 20. PMID 20304396
- [Result] Schouten R, Rijs CS, Bouvy ND, Hameeteman W, Koek GH, Janssen IM, Greve JW. A multicenter, randomized efficacy study of the EndoBarrier Gastrointestinal Liner for presurgical weight loss prior to bariatric surgery. Ann Surg. 2010 Feb;251(2):236-43. doi: 10.1097/SLA.0b013e3181bdfbff. PMID 19858703
- [Result] Escalona A, Pimentel F, Sharp A, Becerra P, Slako M, Turiel D, Munoz R, Bambs C, Guzman S, Ibanez L, Gersin K. Weight loss and metabolic improvement in morbidly obese subjects implanted for 1 year with an endoscopic duodenal-jejunal bypass liner. Ann Surg. 2012 Jun;255(6):1080-5. doi: 10.1097/SLA.0b013e31825498c4. PMID 22534421
- [Result] de Moura EG, Martins BC, Lopes GS, Orso IR, de Oliveira SL, Galvao Neto MP, Santo MA, Sakai P, Ramos AC, Garrido Junior AB, Mancini MC, Halpern A, Cecconello I. Metabolic improvements in obese type 2 diabetes subjects implanted for 1 year with an endoscopically deployed duodenal-jejunal bypass liner. Diabetes Technol Ther. 2012 Feb;14(2):183-9. doi: 10.1089/dia.2011.0152. Epub 2011 Sep 20. PMID 21932999
- [Result] Cohen, R., et al. Endoscopic Duodenal-Jejunal Bypass: Effect on Insulin Sensitivity in Mildly Obese Diabetic Subjects. in 72nd Scientific Sessions American Diabetes Association (Philadelphia, USA, 2012).
- [Result] Mathes CM, Spector AC. Food selection and taste changes in humans after Roux-en-Y gastric bypass surgery: a direct-measures approach. Physiol Behav. 2012 Nov 5;107(4):476-83. doi: 10.1016/j.physbeh.2012.02.013. Epub 2012 Feb 16. PMID 22366157
- [Result] Ochner CN, Kwok Y, Conceicao E, Pantazatos SP, Puma LM, Carnell S, Teixeira J, Hirsch J, Geliebter A. Selective reduction in neural responses to high calorie foods following gastric bypass surgery. Ann Surg. 2011 Mar;253(3):502-7. doi: 10.1097/SLA.0b013e318203a289. PMID 21169809
- [Result] Rodriguez L, Reyes E, Fagalde P, Oltra MS, Saba J, Aylwin CG, Prieto C, Ramos A, Galvao M, Gersin KS, Sorli C. Pilot clinical study of an endoscopic, removable duodenal-jejunal bypass liner for the treatment of type 2 diabetes. Diabetes Technol Ther. 2009 Nov;11(11):725-32. doi: 10.1089/dia.2009.0063. PMID 19905889
- [Result] Escalona A, Yanez R, Pimentel F, Galvao M, Ramos AC, Turiel D, Boza C, Awruch D, Gersin K, Ibanez L. Initial human experience with restrictive duodenal-jejunal bypass liner for treatment of morbid obesity. Surg Obes Relat Dis. 2010 Mar 4;6(2):126-31. doi: 10.1016/j.soard.2009.12.009. Epub 2010 Jan 20. PMID 20359665
- [Result] Breen DM, Rasmussen BA, Kokorovic A, Wang R, Cheung GW, Lam TK. Jejunal nutrient sensing is required for duodenal-jejunal bypass surgery to rapidly lower glucose concentrations in uncontrolled diabetes. Nat Med. 2012 Jun;18(6):950-5. doi: 10.1038/nm.2745. PMID 22610279
- [Result] Thomas C, Pellicciari R, Pruzanski M, Auwerx J, Schoonjans K. Targeting bile-acid signalling for metabolic diseases. Nat Rev Drug Discov. 2008 Aug;7(8):678-93. doi: 10.1038/nrd2619. PMID 18670431
- [Result] Ashrafian H, le Roux CW. Metabolic surgery and gut hormones - a review of bariatric entero-humoral modulation. Physiol Behav. 2009 Jul 14;97(5):620-31. doi: 10.1016/j.physbeh.2009.03.012. Epub 2009 Mar 20. PMID 19303889
- [Result] de Luis D, Domingo M, Romero A, Gonzalez Sagrado M, Pacheco D, Primo D, Conde R. Effects of duodenal-jejunal exclusion on beta cell function and hormonal regulation in Goto-Kakizaki rats. Am J Surg. 2012 Aug;204(2):242-7. doi: 10.1016/j.amjsurg.2011.07.020. Epub 2012 Feb 16. PMID 22341521
- [Result] Speck M, Cho YM, Asadi A, Rubino F, Kieffer TJ. Duodenal-jejunal bypass protects GK rats from beta-cell loss and aggravation of hyperglycemia and increases enteroendocrine cells coexpressing GIP and GLP-1. Am J Physiol Endocrinol Metab. 2011 May;300(5):E923-32. doi: 10.1152/ajpendo.00422.2010. Epub 2011 Feb 8. PMID 21304061
- [Result] Lee HC, Kim MK, Kwon HS, Kim E, Song KH. Early changes in incretin secretion after laparoscopic duodenal-jejunal bypass surgery in type 2 diabetic patients. Obes Surg. 2010 Nov;20(11):1530-5. doi: 10.1007/s11695-010-0248-2. PMID 20803098
- [Result] Kindel TL, Yoder SM, Seeley RJ, D'Alessio DA, Tso P. Duodenal-jejunal exclusion improves glucose tolerance in the diabetic, Goto-Kakizaki rat by a GLP-1 receptor-mediated mechanism. J Gastrointest Surg. 2009 Oct;13(10):1762-72. doi: 10.1007/s11605-009-0912-9. Epub 2009 May 12. PMID 19488823
- [Result] De Silva A, Salem V, Long CJ, Makwana A, Newbould RD, Rabiner EA, Ghatei MA, Bloom SR, Matthews PM, Beaver JD, Dhillo WS. The gut hormones PYY 3-36 and GLP-1 7-36 amide reduce food intake and modulate brain activity in appetite centers in humans. Cell Metab. 2011 Nov 2;14(5):700-6. doi: 10.1016/j.cmet.2011.09.010. Epub 2011 Oct 13. PMID 22000927
- [Result] Dumas ME, Barton RH, Toye A, Cloarec O, Blancher C, Rothwell A, Fearnside J, Tatoud R, Blanc V, Lindon JC, Mitchell SC, Holmes E, McCarthy MI, Scott J, Gauguier D, Nicholson JK. Metabolic profiling reveals a contribution of gut microbiota to fatty liver phenotype in insulin-resistant mice. Proc Natl Acad Sci U S A. 2006 Aug 15;103(33):12511-6. doi: 10.1073/pnas.0601056103. Epub 2006 Aug 8. PMID 16895997
- [Result] Nicholson JK, Holmes E, Wilson ID. Gut microorganisms, mammalian metabolism and personalized health care. Nat Rev Microbiol. 2005 May;3(5):431-8. doi: 10.1038/nrmicro1152. PMID 15821725
- [Result] Williams HR, Cox IJ, Walker DG, North BV, Patel VM, Marshall SE, Jewell DP, Ghosh S, Thomas HJ, Teare JP, Jakobovits S, Zeki S, Welsh KI, Taylor-Robinson SD, Orchard TR. Characterization of inflammatory bowel disease with urinary metabolic profiling. Am J Gastroenterol. 2009 Jun;104(6):1435-44. doi: 10.1038/ajg.2009.175. Epub 2009 Apr 28. PMID 19491857
- [Result] Trygg J, Holmes E, Lundstedt T. Chemometrics in metabonomics. J Proteome Res. 2007 Feb;6(2):469-79. doi: 10.1021/pr060594q. PMID 17269704
- [Result] Calvani R, Miccheli A, Capuani G, Tomassini Miccheli A, Puccetti C, Delfini M, Iaconelli A, Nanni G, Mingrone G. Gut microbiome-derived metabolites characterize a peculiar obese urinary metabotype. Int J Obes (Lond). 2010 Jun;34(6):1095-8. doi: 10.1038/ijo.2010.44. Epub 2010 Mar 9. PMID 20212498
- [Result] Mutch DM, Fuhrmann JC, Rein D, Wiemer JC, Bouillot JL, Poitou C, Clement K. Metabolite profiling identifies candidate markers reflecting the clinical adaptations associated with Roux-en-Y gastric bypass surgery. PLoS One. 2009 Nov 19;4(11):e7905. doi: 10.1371/journal.pone.0007905. PMID 19936240
- [Result] Zhang H, DiBaise JK, Zuccolo A, Kudrna D, Braidotti M, Yu Y, Parameswaran P, Crowell MD, Wing R, Rittmann BE, Krajmalnik-Brown R. Human gut microbiota in obesity and after gastric bypass. Proc Natl Acad Sci U S A. 2009 Feb 17;106(7):2365-70. doi: 10.1073/pnas.0812600106. Epub 2009 Jan 21. PMID 19164560
- [Result] Turnbaugh PJ, Ley RE, Mahowald MA, Magrini V, Mardis ER, Gordon JI. An obesity-associated gut microbiome with increased capacity for energy harvest. Nature. 2006 Dec 21;444(7122):1027-31. doi: 10.1038/nature05414. PMID 17183312
- [Result] Olbers T, Bjorkman S, Lindroos A, Maleckas A, Lonn L, Sjostrom L, Lonroth H. Body composition, dietary intake, and energy expenditure after laparoscopic Roux-en-Y gastric bypass and laparoscopic vertical banded gastroplasty: a randomized clinical trial. Ann Surg. 2006 Nov;244(5):715-22. doi: 10.1097/01.sla.0000218085.25902.f8. PMID 17060764
- [Result] le Roux CW, Bueter M, Theis N, Werling M, Ashrafian H, Lowenstein C, Athanasiou T, Bloom SR, Spector AC, Olbers T, Lutz TA. Gastric bypass reduces fat intake and preference. Am J Physiol Regul Integr Comp Physiol. 2011 Oct;301(4):R1057-66. doi: 10.1152/ajpregu.00139.2011. Epub 2011 Jul 6. PMID 21734019
- [Result] Carey VJ, Walters EE, Colditz GA, Solomon CG, Willett WC, Rosner BA, Speizer FE, Manson JE. Body fat distribution and risk of non-insulin-dependent diabetes mellitus in women. The Nurses' Health Study. Am J Epidemiol. 1997 Apr 1;145(7):614-9. doi: 10.1093/oxfordjournals.aje.a009158. PMID 9098178
- [Result] Manson JE, Colditz GA, Stampfer MJ, Willett WC, Rosner B, Monson RR, Speizer FE, Hennekens CH. A prospective study of obesity and risk of coronary heart disease in women. N Engl J Med. 1990 Mar 29;322(13):882-9. doi: 10.1056/NEJM199003293221303. PMID 2314422
- [Result] Calle EE, Thun MJ, Petrelli JM, Rodriguez C, Heath CW Jr. Body-mass index and mortality in a prospective cohort of U.S. adults. N Engl J Med. 1999 Oct 7;341(15):1097-105. doi: 10.1056/NEJM199910073411501. PMID 10511607
- [Result] Rao Kondapally Seshasai S, Kaptoge S, Thompson A, Di Angelantonio E, Gao P, Sarwar N, Whincup PH, Mukamal KJ, Gillum RF, Holme I, Njolstad I, Fletcher A, Nilsson P, Lewington S, Collins R, Gudnason V, Thompson SG, Sattar N, Selvin E, Hu FB, Danesh J; Emerging Risk Factors Collaboration. Diabetes mellitus, fasting glucose, and risk of cause-specific death. N Engl J Med. 2011 Mar 3;364(9):829-841. doi: 10.1056/NEJMoa1008862. PMID 21366474
- [Result] American Diabetes Association. Standards of medical care in diabetes--2013. Diabetes Care. 2013 Jan;36 Suppl 1(Suppl 1):S11-66. doi: 10.2337/dc13-S011. No abstract available. PMID 23264422
- [Result] Oldfield RC. The assessment and analysis of handedness: the Edinburgh inventory. Neuropsychologia. 1971 Mar;9(1):97-113. doi: 10.1016/0028-3932(71)90067-4. No abstract available. PMID 5146491
- [Result] Inzucchi SE, Bergenstal RM, Buse JB, Diamant M, Ferrannini E, Nauck M, Peters AL, Tsapas A, Wender R, Matthews DR; American Diabetes Association (ADA); European Association for the Study of Diabetes (EASD). Management of hyperglycemia in type 2 diabetes: a patient-centered approach: position statement of the American Diabetes Association (ADA) and the European Association for the Study of Diabetes (EASD). Diabetes Care. 2012 Jun;35(6):1364-79. doi: 10.2337/dc12-0413. Epub 2012 Apr 19. No abstract available. PMID 22517736
- [Result] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Result] Rankinen T, Bouchard C. Genetics of food intake and eating behavior phenotypes in humans. Annu Rev Nutr. 2006;26:413-34. doi: 10.1146/annurev.nutr.26.061505.111218. PMID 16848714
- [Result] Bell CG, Walley AJ, Froguel P. The genetics of human obesity. Nat Rev Genet. 2005 Mar;6(3):221-34. doi: 10.1038/nrg1556. PMID 15703762
- [Result] Miller FA, Ahern C, Smith CA, Harvey EA. Understanding the new human genetics: a review of scientific editorials. Soc Sci Med. 2006 May;62(10):2373-85. doi: 10.1016/j.socscimed.2005.11.015. Epub 2005 Dec 27. PMID 16377046
- [Result] van Strien, T., Frijters, J.E.R., Bergers, G.P.A. & Defares, P.B. The Dutch Eating Behavior Questionnaire (DEBQ) for assessment of restrained, emotional, and external eating behavior. Int J Eat Disorder 5, 295-315 (1986).
- [Result] Kroke A, Klipstein-Grobusch K, Voss S, Moseneder J, Thielecke F, Noack R, Boeing H. Validation of a self-administered food-frequency questionnaire administered in the European Prospective Investigation into Cancer and Nutrition (EPIC) Study: comparison of energy, protein, and macronutrient intakes estimated with the doubly labeled water, urinary nitrogen, and repeated 24-h dietary recall methods. Am J Clin Nutr. 1999 Oct;70(4):439-47. doi: 10.1093/ajcn/70.4.439. PMID 10500011
- [Result] Patton JH, Stanford MS, Barratt ES. Factor structure of the Barratt impulsiveness scale. J Clin Psychol. 1995 Nov;51(6):768-74. doi: 10.1002/1097-4679(199511)51:63.0.co;2-1. PMID 8778124
- [Result] Yeomans MR, Leitch M, Mobini S. Impulsivity is associated with the disinhibition but not restraint factor from the Three Factor Eating Questionnaire. Appetite. 2008 Mar-May;50(2-3):469-76. doi: 10.1016/j.appet.2007.10.002. Epub 2007 Oct 18. PMID 18069081
- [Result] Heatherton TF, Kozlowski LT, Frecker RC, Fagerstrom KO. The Fagerstrom Test for Nicotine Dependence: a revision of the Fagerstrom Tolerance Questionnaire. Br J Addict. 1991 Sep;86(9):1119-27. doi: 10.1111/j.1360-0443.1991.tb01879.x. PMID 1932883
- [Result] Stunkard AJ, Messick S. The three-factor eating questionnaire to measure dietary restraint, disinhibition and hunger. J Psychosom Res. 1985;29(1):71-83. doi: 10.1016/0022-3999(85)90010-8. PMID 3981480
- [Result] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865
- [Result] Killgore WD, Yurgelun-Todd DA. Affect modulates appetite-related brain activity to images of food. Int J Eat Disord. 2006 Jul;39(5):357-63. doi: 10.1002/eat.20240. PMID 16565998
- [Result] Gearhardt AN, Corbin WR, Brownell KD. Preliminary validation of the Yale Food Addiction Scale. Appetite. 2009 Apr;52(2):430-6. doi: 10.1016/j.appet.2008.12.003. Epub 2008 Dec 11. PMID 19121351
- [Result] Babor, T., Higgins-Biddle, J., Saunders, J. & Monteiro, M. AUDIT: The Alcohol Use Disorders Identification Test: Guidelines for Use in Primary Care. (2001).
- [Result] Lowe MR, Butryn ML, Didie ER, Annunziato RA, Thomas JG, Crerand CE, Ochner CN, Coletta MC, Bellace D, Wallaert M, Halford J. The Power of Food Scale. A new measure of the psychological influence of the food environment. Appetite. 2009 Aug;53(1):114-8. doi: 10.1016/j.appet.2009.05.016. Epub 2009 Jun 12. PMID 19500623
- [Result] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Result] Sigstad H. A clinical diagnostic index in the diagnosis of the dumping syndrome. Changes in plasma volume and blood sugar after a test meal. Acta Med Scand. 1970 Dec;188(6):479-86. No abstract available. PMID 5507449
- [Result] Arts J, Caenepeel P, Bisschops R, Dewulf D, Holvoet L, Piessevaux H, Bourgeois S, Sifrim D, Janssens J, Tack J. Efficacy of the long-acting repeatable formulation of the somatostatin analogue octreotide in postoperative dumping. Clin Gastroenterol Hepatol. 2009 Apr;7(4):432-7. doi: 10.1016/j.cgh.2008.11.025. Epub 2008 Dec 13. PMID 19264574
- [Result] Gormally J, Black S, Daston S, Rardin D. The assessment of binge eating severity among obese persons. Addict Behav. 1982;7(1):47-55. doi: 10.1016/0306-4603(82)90024-7. PMID 7080884
- [Result] Herrmann C. Screening for major depression in a group of diabetic patients. Psychosom Med. 1997 Sep-Oct;59(5):559-60. doi: 10.1097/00006842-199709000-00016. No abstract available. PMID 9316191
- [Result] Stewart AL, Hays RD, Ware JE Jr. The MOS short-form general health survey. Reliability and validity in a patient population. Med Care. 1988 Jul;26(7):724-35. doi: 10.1097/00005650-198807000-00007. No abstract available. PMID 3393032
- [Result] Kirby KN, Marakovic NN. Delay-discounting probabilistic rewards: Rates decrease as amounts increase. Psychon Bull Rev. 1996 Mar;3(1):100-4. doi: 10.3758/BF03210748. PMID 24214810
- [Result] Kirby KN, Petry NM. Heroin and cocaine abusers have higher discount rates for delayed rewards than alcoholics or non-drug-using controls. Addiction. 2004 Apr;99(4):461-71. doi: 10.1111/j.1360-0443.2003.00669.x. PMID 15049746
- [Result] Perry JL, Carroll ME. The role of impulsive behavior in drug abuse. Psychopharmacology (Berl). 2008 Sep;200(1):1-26. doi: 10.1007/s00213-008-1173-0. Epub 2008 Jul 5. PMID 18600315
- [Result] Weller RE, Cook EW 3rd, Avsar KB, Cox JE. Obese women show greater delay discounting than healthy-weight women. Appetite. 2008 Nov;51(3):563-9. doi: 10.1016/j.appet.2008.04.010. Epub 2008 Apr 18. PMID 18513828
- [Result] Davis C, Patte K, Curtis C, Reid C. Immediate pleasures and future consequences. A neuropsychological study of binge eating and obesity. Appetite. 2010 Feb;54(1):208-13. doi: 10.1016/j.appet.2009.11.002. Epub 2009 Nov 5. PMID 19896515
- [Result] Finlayson G, King N, Blundell J. The role of implicit wanting in relation to explicit liking and wanting for food: implications for appetite control. Appetite. 2008 Jan;50(1):120-7. doi: 10.1016/j.appet.2007.06.007. Epub 2007 Jun 28. PMID 17655972
- [Result] Haidt, J., Mccauley, C. & Rozin, P. Individual-Differences in Sensitivity to Disgust - a Scale Sampling 7 Domains of Disgust Elicitors. Pers Indiv Differ 16, 701-713 (1994).
- [Result] Olatunji BO, Williams NL, Tolin DF, Abramowitz JS, Sawchuk CN, Lohr JM, Elwood LS. The Disgust Scale: item analysis, factor structure, and suggestions for refinement. Psychol Assess. 2007 Sep;19(3):281-97. doi: 10.1037/1040-3590.19.3.281. PMID 17845120
- [Result] Petersen ET, Zimine I, Ho YC, Golay X. Non-invasive measurement of perfusion: a critical review of arterial spin labelling techniques. Br J Radiol. 2006 Aug;79(944):688-701. doi: 10.1259/bjr/67705974. PMID 16861326
- [Result] Paiva FF, Tannus A, Silva AC. Measurement of cerebral perfusion territories using arterial spin labelling. NMR Biomed. 2007 Nov;20(7):633-42. doi: 10.1002/nbm.1177. PMID 17503440
- [Result] Damoiseaux JS, Rombouts SA, Barkhof F, Scheltens P, Stam CJ, Smith SM, Beckmann CF. Consistent resting-state networks across healthy subjects. Proc Natl Acad Sci U S A. 2006 Sep 12;103(37):13848-53. doi: 10.1073/pnas.0601417103. Epub 2006 Aug 31. PMID 16945915
- [Result] Goldstone AP, Prechtl de Hernandez CG, Beaver JD, Muhammed K, Croese C, Bell G, Durighel G, Hughes E, Waldman AD, Frost G, Bell JD. Fasting biases brain reward systems towards high-calorie foods. Eur J Neurosci. 2009 Oct;30(8):1625-35. doi: 10.1111/j.1460-9568.2009.06949.x. Epub 2009 Oct 7. PMID 19811532
- [Result] Knutson B, Adams CM, Fong GW, Hommer D. Anticipation of increasing monetary reward selectively recruits nucleus accumbens. J Neurosci. 2001 Aug 15;21(16):RC159. doi: 10.1523/JNEUROSCI.21-16-j0002.2001. PMID 11459880
- [Result] Knutson B, Westdorp A, Kaiser E, Hommer D. FMRI visualization of brain activity during a monetary incentive delay task. Neuroimage. 2000 Jul;12(1):20-7. doi: 10.1006/nimg.2000.0593. PMID 10875899
- [Result] Li CS, Yan P, Chao HH, Sinha R, Paliwal P, Constable RT, Zhang S, Lee TW. Error-specific medial cortical and subcortical activity during the stop signal task: a functional magnetic resonance imaging study. Neuroscience. 2008 Sep 9;155(4):1142-51. doi: 10.1016/j.neuroscience.2008.06.062. Epub 2008 Jul 8. PMID 18674592
- [Result] Berger S. The WAIS-R factors: usefulness and construct validity in neuropsychological assessments. Appl Neuropsychol. 1998;5(1):37-42. doi: 10.1207/s15324826an0501_5. PMID 16318465
- [Result] Bueter M, Miras AD, Chichger H, Fenske W, Ghatei MA, Bloom SR, Unwin RJ, Lutz TA, Spector AC, le Roux CW. Alterations of sucrose preference after Roux-en-Y gastric bypass. Physiol Behav. 2011 Oct 24;104(5):709-21. doi: 10.1016/j.physbeh.2011.07.025. Epub 2011 Jul 30. PMID 21827777
- [Result] Dixon JB, Zimmet P, Alberti KG, Rubino F; International Diabetes Federation Taskforce on Epidemiology and Prevention. Bariatric surgery: an IDF statement for obese Type 2 diabetes. Diabet Med. 2011 Jun;28(6):628-42. doi: 10.1111/j.1464-5491.2011.03306.x. PMID 21480973
- [Result] Gaede P, Lund-Andersen H, Parving HH, Pedersen O. Effect of a multifactorial intervention on mortality in type 2 diabetes. N Engl J Med. 2008 Feb 7;358(6):580-91. doi: 10.1056/NEJMoa0706245. PMID 18256393
- [Result] Philips Z, Ginnelly L, Sculpher M, Claxton K, Golder S, Riemsma R, Woolacoot N, Glanville J. Review of guidelines for good practice in decision-analytic modelling in health technology assessment. Health Technol Assess. 2004 Sep;8(36):iii-iv, ix-xi, 1-158. doi: 10.3310/hta8360. PMID 15361314
- [Result] Caro JJ, Briggs AH, Siebert U, Kuntz KM; ISPOR-SMDM Modeling Good Research Practices Task Force. Modeling good research practices--overview: a report of the ISPOR-SMDM Modeling Good Research Practices Task Force-1. Med Decis Making. 2012 Sep-Oct;32(5):667-77. doi: 10.1177/0272989X12454577. PMID 22990082
- [Result] Mount Hood 4 Modeling Group. Computer modeling of diabetes and its complications: a report on the Fourth Mount Hood Challenge Meeting. Diabetes Care. 2007 Jun;30(6):1638-46. doi: 10.2337/dc07-9919. PMID 17526823
- [Result] Stevens RJ, Kothari V, Adler AI, Stratton IM; United Kingdom Prospective Diabetes Study (UKPDS) Group. The UKPDS risk engine: a model for the risk of coronary heart disease in Type II diabetes (UKPDS 56). Clin Sci (Lond). 2001 Dec;101(6):671-9. PMID 11724655
- [Result] Clarke P, Gray A, Holman R. Estimating utility values for health states of type 2 diabetic patients using the EQ-5D (UKPDS 62). Med Decis Making. 2002 Jul-Aug;22(4):340-9. doi: 10.1177/0272989X0202200412. PMID 12150599
- [Derived] Glaysher MA, Ward J, Aldhwayan M, Ruban A, Prechtl CG, Fisk HL, Chhina N, Al-Najim W, Smith C, Klimowska-Nassar N, Johnson N, Falaschetti E, Goldstone AP, Miras AD, Byrne JP, Calder PC, Teare JP. The effect of a duodenal-jejunal bypass liner on lipid profile and blood concentrations of long chain polyunsaturated fatty acids. Clin Nutr. 2021 Apr;40(4):2343-2354. doi: 10.1016/j.clnu.2020.10.026. Epub 2020 Oct 22. PMID 33131909
- [Derived] Glaysher MA, Mohanaruban A, Prechtl CG, Goldstone AP, Miras AD, Lord J, Chhina N, Falaschetti E, Johnson NA, Al-Najim W, Smith C, Li JV, Patel M, Ahmed AR, Moore M, Poulter N, Bloom S, Darzi A, Le Roux C, Byrne JP, Teare JP. A randomised controlled trial of a duodenal-jejunal bypass sleeve device (EndoBarrier) compared with standard medical therapy for the management of obese subjects with type 2 diabetes mellitus. BMJ Open. 2017 Nov 15;7(11):e018598. doi: 10.1136/bmjopen-2017-018598. PMID 29146657
- See also: Official Trial Website — http://www1.imperial.ac.uk/biosurgerysurgicaltechnology/clinical_trials_outcomes/bariatricsurgery/endobarrier/